CLINICAL TRIAL: NCT07177716
Title: A Multicenter, Randomized, Open-Label Phase II/III Clinical Study on the Efficacy and Safety of LB1410 Plus Lenvatinib With or Without LB4330 Versus Investigator's Choice of Chemotherapy in Advanced Recurrent/Metastatic Cervical Cancer
Brief Title: Efficacy and Safety of LB1410 Plus Lenvatinib With or Without LB4330 in Advanced Recurrent/Metastatic Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: L & L Bio Co., Ltd., Ningbo, China (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LB1410-CC01
Record Dates: First submitted 2025-09-04; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer
Keywords: cervical carcinoma; LB1410; LB4330
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: LB1410 + Lenvatinib (Experimental): LB1410 (intravenous, Q2W) with lenvatinib (oral, QD),up to 2 years
  Interventions: Biological: LB1410; Drug: Lenvatinib
- Cohort 2: LB1410 + LB4330 + Lenvatinib (Experimental): LB1410 (IV, Q2W for up to 2 years), LB4330 (IV, Q2W for 4 cycles), and lenvatinib (oral, once daily for up to 2 years)
  Interventions: Biological: LB1410; Biological: LB4330; Drug: Lenvatinib
- Cohort 3: LB1410 (Experimental): LB1410 (IV, Q2W for up to 2 years)
  Interventions: Biological: LB1410
- Cohort 4: LB1410 + LB4330 (Experimental): LB1410 (IV, Q2W for up to 2 years) plus LB4330 (IV, Q2W for 4 cycles)
  Interventions: Biological: LB1410; Biological: LB4330

INTERVENTIONS:
Biological: LB1410 — LB1410 (IV, Q2W for up to 2 years)
Biological: LB4330 — LB4330 (IV, Q2W for 4 cycles)
  Arms: Cohort 2: LB1410 + LB4330 + Lenvatinib; Cohort 4: LB1410 + LB4330
Drug: Lenvatinib — lenvatinib (oral, once daily for up to 2 years)
  Arms: Cohort 1: LB1410 + Lenvatinib; Cohort 2: LB1410 + LB4330 + Lenvatinib

SUMMARY:
This is a multicenter, randomized, open-label Phase II/III clinical study, aiming to evaluate the efficacy and safety of LB1410 in combination with lenvatinib (whether in combination with LB4330）versus the chemotherapy regimen selected by the investigators for patients with advanced recurrent/metastatic cervical cancer.

DETAILED DESCRIPTION:
This study is an open-label, multicenter Phase II/III clinical trial in advanced/metastatic cervical cancer to evaluate the antitumor efficacy, safety, tolerability, pharmacokinetics (PK), and biomarkers of LB1410 in combination with lenvatinib, with or without LB4330.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed cervical squamous cell carcinoma, adenosquamous carcinoma, or HPV-associated cervical adenocarcinoma.
2. Recurrent or metastatic cervical cancer with disease progression or intolerable toxicity after standard therapy, with no more than three prior lines of systemic therapy in the recurrent or metastatic setting, with only one prior line of therapy containing anti-PD-1/anti-PD-L1 agents.
3. At least one measurable lesion per RECIST v1.1 at screening period.
4. Age ≥18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Investigator-assessed life expectancy ≥12 weeks.
7. Adequate hematological function, liver function, renal function and coagulation function.
8. Adequately controlled blood pressure (BP) with or without antihypertensive medication.
9. Any related toxicity or prior adverse events (AEs) had recovered to baseline or ≤Grade 1 per NCI CTCAE v5.0.
10. Women of childbearing potential must agree to use effective contraception from the time of signing the informed consent form, throughout the study, and for 6 months after the last dose of study treatment.
11. The patient is capable of understanding and voluntarily signing the informed consent form.

Exclusion Criteria

1. For cohorts containing lenvatinib, patients meeting any of the following criteria are ineligible:

   1. Radiographic (CT or MRI) evidence of tumor invasion around major blood vessels, or investigator judgment that the tumor is highly likely to invade major blood vessels during the study, leading to life-threatening hemorrhage;
   2. History of bleeding, coagulation disorders, or current use of warfarin, aspirin, or other antiplatelet agents;
   3. Urine protein ≥2+ and 24-hour urine protein quantification ≥1.0 g;
   4. Factors affecting oral drug absorption;
   5. Intestinal metastases or existing ≥Grade 3 gastrointestinal or non-gastrointestinal fistulas;
   6. History of hypertensive crisis or hypertensive encephalopathy.
2. Pregnant or breastfeeding women.
3. History of ≥Grade 3 immune-related adverse events (irAEs) during prior immunotherapy.
4. Active autoimmune disease or symptomatic autoimmune disease.
5. Any of the following prior treatments:

   1. Live or attenuated live vaccines within 4 weeks before the first dose;
   2. Immunomodulatory drugs (e.g., thymosin, interleukin-2, interferon) within 14 days before the first dose;
   3. History of allogeneic organ transplantation, allogeneic peripheral hematopoietic stem cell transplantation, or bone marrow transplantation.
6. Positive HIV test, active syphilis, active hepatitis B virus (HBV) infection, or active hepatitis C virus (HCV) infection.
7. Other malignancies within the past 3 year.
8. Leptomeningeal metastasis, spinal cord compression, symptomatic or unstable brain metastases.
9. Uncontrolled or poorly controlled diabetes.
10. Arterial/venous thrombotic events within 6 months.
11. Clinically significant and unstable pleural, peritoneal, or pericardial effusion.
12. Known interstitial lung disease.
13. Prior use of drugs with the same mechanism as this study (e.g., PD-1 antibody combined with TIM-3 antibody, PD-1/TIM-3 bispecific antibodies).
14. Any other condition (including severe medical or psychiatric illness) or clinically significant laboratory abnormality that may affect patient safety or study integrity per investigator judgment.
15. (Applicable only to containing-LB4330 cohorts): History of Grade IV thrombocytopenia (per CTCAE) from any prior anti-cancer regimen within the past 2 years, or prior exposure to any interleukin-10 (IL-10) based agent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assessed by an Independent Radiology Review Committee (IRRC) | Approximately 24 months
  defined as the percentage of patients with a best overall response of Complete Response or Partial Response per RECIST 1.1.
Duration of Response (DOR) assessed by an Independent Radiology Review Committee (IRRC) | Approximately 24 months
  defined as the time from the first documented response (CR or PR) to the first documented disease progression or death due to underlying cancer per RECIST 1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) assessed by the investigator | Approximately 24 months
  defined as the percentage of patients with a best overall response of Complete Response or Partial Response per RECIST 1.1.
Duration of Response (DOR) assessed by the investigator | Approximately 24 months
  defined as the time from the first documented response (CR or PR) to the first documented disease progression or death due to underlying cancer per RECIST 1.1.
Disease Control Rate (DCR) | Approximately 24 months
  defined as the percentage of evaluable patients achieving a best overall response of complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1 assessed by both the investigator and an Independent Radiology Review Committee (IRRC).
Progression-Free Survival (PFS) | Approximately 24 months
  defined as the time from the first dose to the first documented disease progression per RECIST 1.1 or death due to any cause (whichever occurred first) assessed by both the investigator and an IRRC.
Overall Survival (OS) | Until participant death/end of study,approximately 24 months
  Overall Survival is defined as the time from the date of first study treatment to the date of death from any cause or the date of censoring.
Safety and tolerability (Adverse Event reported per NCI-CTCAE v5.0) | From the first dose administration to 30 days after the last dose
  Incidence of treatment-emergent adverse events (TEAEs) and treatment-related adverse events reported per NCI-CTCAE v5.0
ADA Antibody Positivity Rate of LB1410 | From the first dose administration to 30 days after the last dose
  ADA Antibody Positivity Rate of LB1410
Pharmacokinetic (PK) parameters of LB1410-Maximum (peak) Plasma Concentration（Cmax） | From the first dose administration to Cycle 16 Day 1 (each cycle is 28 days)
  The highest concentration a drug reaches in the bloodstream after a single dose.
Pharmacokinetic (PK) parameters of LB1410-Trough Concentration（Ctrough） | From the first dose administration to Cycle 16 Day 1 (each cycle is 28 days)
  The minimum drug concentration at steady state, measured just before the next dose is administered.
Pharmacokinetic (PK) parameters of LB1410-Area Under the Curve at Steady State(AUCss) | From the first dose administration to Cycle 16 Day 1 (each cycle is 28 days)
  The total area under the plasma concentration-time curve over one dosing interval at steady state, representing total drug exposure.

OTHER OUTCOMES:
Biomarker(TIM3) | Until end of study,approximately 24 months
  Correlation between TIM3 expression and clinical efficacy endpoints (ORR, DCR, PFS, OS) as assessed by the investigator according to RECIST 1.1 criteria.
Biomarker(PD-L1) | Until end of study,approximately 24 months
  Correlation between PD-L1 expression and clinical efficacy endpoints (ORR, DCR, PFS, OS) as assessed by the investigator according to RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No